CLINICAL TRIAL: NCT06290947
Title: Evaluating the Impact of Blood-Flow Restriction Walk Training on Insulin Sensitivity and Aerobic Capacity in Individuals With Type 2 Diabetes Mellitus: A Randomized Controlled Trial
Brief Title: BFR Walking for Insulin and Aerobic Improvement in Type 2 Diabetes
Acronym: BRAID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arab American University (Palestine) (Other)
Responsible Party: Principal Investigator, Samer AbuEid, Assistant Professor, Arab American University (Palestine)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: BFR-AE-DT2-2023-01; IRB 2022/C/20/N (Other Grant/Funding Number: AAUP)
Record Dates: First submitted 2024-02-21; First posted 2024-03-04 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-03

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes Mellitus; Blood-Flow Restriction Training (BFR); Insulin Sensitivity; Aerobic Capacity; Diabetes Management; Low-Intensity Exercise
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance

STUDY DESIGN:
Intervention Model Description: This study employs a randomized controlled trial model with a parallel assignment to evaluate the efficacy of Blood-Flow Restriction Walk Training compared to a control condition. Participants are randomly allocated into two groups: one receiving the intervention (BFR walk training) and the other serving as a control (usual walk training). This design allows for the direct comparison of outcomes between the intervention and control groups over the study period.
Masking Description: None (Open Label)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Blood-Flow Restriction Walk Training (BFRw) (Experimental): Participants in this group will engage in a Blood-Flow Restriction Walk Training (BFRw) program designed to evaluate the efficacy of BFRw in enhancing insulin sensitivity and aerobic capacity.
  Activities:
  Participants will attend three weekly supervised walking sessions for eight weeks, each integrating specialized BFR cuffs calibrated to a precise pressure to restrict blood flow during exercise partially.
  Purpose:
  This arm is crucial for testing the study's primary hypothesis by measuring the intervention's effects against a control group.
  Interventions: Device: BFR Cuffs for Intervention Group; Other: Standard Walking Training Program
- Control Group Walk Training (Active Comparator): Participants in this group will engage in a conventional walking training program without applying BFR cuffs.
  Activities:
  Participants will attend three weekly supervised walking sessions for eight weeks without using BFR cuffs.
  Purpose:
  This group will serve as a benchmark to ascertain the effectiveness of the intervention, providing a baseline for the comparative analysis of the results obtained from the intervention group.
  Interventions: Other: Standard Walking Training Program

INTERVENTIONS:
Device: BFR Cuffs for Intervention Group — The intervention consists of supervised treadmill sessions incorporating specialized BFR cuffs, branded as "H+ Curve," tailored for Blood-Flow Restriction Walk Training (BFRw). These cuffs are strategically positioned on the upper portion of the lower limbs to induce muscle adaptations and
  improve metabolic health outcomes. The innovative protocol is designed to probe the potential benefits of BFRw in ameliorating insulin sensitivity and enhancing aerobic capacity, thus presenting a pioneering exercise approach for individuals with Type 2 Diabetes.
  Other Names: H+ Cuff 2.0 CURVED BFR Cuffs
  Arms: Blood-Flow Restriction Walk Training (BFRw)
Other: Standard Walking Training Program — The control group will engage in a standard walking training regimen, consisting of supervised treadmill sessions without the application of BFR cuffs. This protocol serves to uphold the scientific rigor of the study by offering a comparison group for the BFRw intervention.
  Purpose:
  To evaluate the impact of a typical exercise routine on insulin sensitivity and aerobic capacity, thereby establishing a control benchmark to contrast with the effects of the BFRw intervention.

SUMMARY:
This clinical trial examines the impact of Blood-Flow Restriction Walk Training (BFRw) on insulin sensitivity and aerobic capacity in individuals with Type 2 Diabetes (T2D).

The primary objectives of the study are to determine: If Blood-Flow Restriction Walk Training (BFRw) can improve insulin sensitivity in individuals with Type 2 Diabetes (T2D).

Whether Blood-Flow Restriction Walk Training (BFRw) enhances aerobic capacity in individuals with Type 2 Diabetes (T2D).

Participants in the study are divided into two groups. One group undergoes Blood-Flow Restriction Walk Training (BFRw), and the other serves as a control. Both groups attend three treadmill walking sessions weekly for eight weeks. The BFRw group has a restriction cuff placed around both thighs during their sessions, while the control group participates in the walking sessions without any blood flow restriction.

Hemoglobin A1c (HbA1c) levels and maximal oxygen consumption (VO2 max) are monitored as indicators of insulin sensitivity and aerobic capacity, respectively.

DETAILED DESCRIPTION:
In this clinical trial, the efficacy of Blood-Flow Restriction Walk Training (BFRw) as a therapeutic modality to enhance insulin sensitivity and aerobic capacity is meticulously explored among individuals diagnosed with Type 2 Diabetes. This innovative approach combines the simplicity of low-intensity walking exercises with the physiological benefits of blood-flow restriction applied to the lower extremities, proposing that such a combination can induce muscle adaptations typically associated with high-intensity resistance training.

The study is centered around a rigorously structured protocol, in which participants assigned to the intervention arm undergo supervised BFRw sessions. These sessions are carefully calibrated to ensure a balance between safety and effectiveness, with a focus on gradually increasing the intensity and duration of the exercise to accommodate the varying fitness levels of participants and to mitigate any potential risks associated with blood-flow restriction techniques.

The research primarily investigates the hypothesis that BFRw can lead to significant improvements in metabolic health markers and physical performance metrics without the physical strain associated with traditional high-intensity exercise regimes. By examining the incremental adaptation of skeletal muscle under conditions of reduced oxygen supply, the study aims to uncover the mechanisms through which BFRw supports enhancements in glucose metabolism and cardiovascular fitness.

Furthermore, the study seeks to identify the optimal parameters for blood-flow restriction that maximize therapeutic benefits while minimizing discomfort and potential complications. This involves comprehensive assessments of insulin sensitivity (via glucose tolerance tests and insulin assays) and aerobic capacity (measured through graded exercise testing to determine VO2 max).

This investigation is designed to provide valuable insights into the feasibility, safety, and efficacy of incorporating Blood-Flow Restriction Walk Training into the treatment regimen for Type 2 Diabetes. By redefining exercise recommendations for individuals with limited tolerance for traditional high-intensity workouts, the research could significantly impact future guidelines and practices for managing this prevalent metabolic disorder.

ELIGIBILITY:
Inclusion Criteria:

* Male individuals of Palestinian descent
* Aged between 40 to 65 years
* Diagnosed with Type 2 Diabetes for a duration of 2 to 10 years, with ongoing medical supervision
* Capable of understanding and following the study's instructions, programs, and protocols

Exclusion Criteria:

* Females, due to hormonal and metabolic differences.
* Individuals outside the 40-65 age range to minimize age-related variations in Diabetes Mellitus.
* Patients with conditions or comorbidities that impair walking or elevate the risk associated with Blood-Flow Restriction Training (BFRT).
* An Ankle Brachial Pressure Index (ABI) greater than 0.9, as values outside the normal range (0.9 to 1.4) may indicate Peripheral Arterial Disease (PAD) or Cardiovascular Disease (CVD), affecting eligibility for participation.

Ages: 40 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-03-06 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2024-01-08 (Actual)

PRIMARY OUTCOMES:
Improvement in Insulin Sensitivity | 8 weeks
  This measure assesses the change in insulin sensitivity determined by cumulative sugar measure.
Improvement in Aerobic Capacity | 8 weeks
  This outcome measure will evaluate the change in aerobic capacity as indicated by VO2 max (maximal oxygen consumption) levels. This assessment will determine the effectiveness of Blood-Flow Restriction Walk Training in enhancing aerobic efficiency in participants.

SECONDARY OUTCOMES:
Change in Body Mass Index (BMI) | 8 weeks
  This outcome will track the change in participants' Body Mass Index (BMI) to assess any impact of Blood-Flow Restriction Walk Training on body composition. BMI will be calculated using measured weight and height at baseline and at the end of the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Samer AbuEid, PhD, Principal Investigator
Locations (1):
- Arab American University - Palestine, Jenin, Palestinian Territories

IPD SHARING:
Plan to Share IPD: No